CLINICAL TRIAL: NCT05523726
Title: Preventing Insomnia and Depression With Nurse Coaching in Individuals With Low Socioeconomic Position
Brief Title: Preventing Insomnia With Virtual Oneshot Therapy (PIVOT)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Philip Cheng, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15827-07
Record Dates: First submitted 2022-08-25; First posted 2022-08-31 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Insomnia
Keywords: Insomnia; Depression; Digital Nurse Coaching; CBT-I; preventative therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Random assignment into experimental and control conditions at a 1:1 ratio
Who Masked: Investigator
Masking Description: The principle investigator will be blind to the group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preventative Cognitive Behavioral Therapy for Insomnia (Experimental): Participants in this group will complete daily sleep diary entries for one week, and then have a telehealth pCBT-I session with a nurse coach, where they will receive personalized sleep recommendations to improve sleep quality.
  Interventions: Behavioral: pCBT-I
- Digital Sleep Education Control (No Intervention): Participants in this group will receive digital sleep education, including tips on how to improve your sleep via interactive email. These materials are selected to help prevent chronic insomnia.

INTERVENTIONS:
Behavioral: pCBT-I — Telehealth coaching
  Arms: Preventative Cognitive Behavioral Therapy for Insomnia

SUMMARY:
This study is intended to assess the efficacy of preventative Cognitive Behavioral Therapy for Insomnia (pCBT-I) on reducing the severity and stopping the progression of acute insomnia and depression. We also hope to gain a deeper understanding of the sociocultural, interpersonal, and individual factors that may have a role in development of insomnia and/or engagement with treatment plans.

DETAILED DESCRIPTION:
Insomnia is a debilitating condition that escalates the risk of a myriad of disorders and is a source of significant economic burden. Insomnia takes an immense toll on individuals' physical and mental wellbeing and treating it before it can develop into chronic insomnia can save individuals untold time and money on treatment.

This study is intended to assess the effects of one virtual pCBT-I session with a nurse coach on reducing the severity and stopping the progression of acute insomnia and depression. The benefits of pCBT-I have been demonstrated in prior studies but have yet to be tested on larger sample populations.

Participants will be recruited from the Henry Ford Health System (HFHS) outpatient network, as well as the Medicare/Medicaid data warehouse and other community partners. Subjects will be screened to determine eligibility, and then will be randomized into one of two insomnia treatment groups (control digital sleep education and pCBT-I via telehealth coaching).

Upon completion, the proposed research will not only have validated a preventative treatment for both insomnia and depression, but we will have the tools to apply it in the most effective way possible.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with low socioeconomic position as defined by income (<35k annual household income) or education (high school diploma or less)
* Experiencing symptoms of prodromal acute insomnia (difficulty falling asleep, difficulty staying asleep, or problems waking up too early), along with worry or distress regarding their symptoms.

Exclusion Criteria:

* Under the age of 18
* Unwilling/unable to participate
* Conditions that could interfere with pCBT-I (including bipolar and seizure disorders)
* Untreated sleep disorders besides insomnia (e.g., sleep apnea, narcolepsy)
* Untreated and severe medical or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity | up to one year post-treatment
  Insomnia Severity Index Score (0 to 28; higher scores correspond to worse severity)
Depression Severity | up to one year post-treatment
  QIDS-SR16 Score (0-27; higher scores correspond to worse severity)
Cases of DSM-5 Insomnia | 6 months post-treatment
  Meet all DSM-5 criteria for Chronic Insomnia
Cases of Clinically Significant Depression | 6-months post-treatment
  QIDS-SR16 score of 11 or higher

SECONDARY OUTCOMES:
Physical Environment | Through study completion, an average of 1 year
  Participants will be asked about the layout of their sleep environment as well as neighborhood characteristics. Sleep environment will be assessed using qualitative information on individual's surroundings and information such as their ability to adjust light levels, temperature, and sound. If it is easier for the individual to adjust these, then they have a better physical environment for sleep. Neighborhood characteristics will be evaluated with the Neighborhood Safety scale (scores range from 1 to 5; lower scores indicate more neighborhood safety).
Sociocultural Environment | Through study completion, an average of 1 year
  Sociocultural environment is measured using a household roster and the Everyday Discrimination Scale. A household roster will ask participants to report the number of individuals in the household and characterize the relationship with the participant. No summary score exists for the household roster. The Everyday Discrimination Scale measures frequency of discrimination (scores range from 10 to 60; higher scores represent more frequent experiences of discrimination).

CONTACTS AND LOCATIONS:
Overall Officials: Philip Cheng, Ph.D., Principal Investigator — Henry Ford Health
Locations (1):
- Henry Ford Columbus Medical Center, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: No